CLINICAL TRIAL: NCT04810637
Title: A Phase 2, Randomized, Double Blinded, Placebo Controlled, Parallel Group, Single Administration Study to Evaluate the Safety and Efficacy of GX-I7 in Elderly Patients With Asymptomatic or Mild Symptoms of COVID-19
Brief Title: A Study to Evaluate the Safety and Efficacy of GX-I7 in Elderly Patients With Asymptomatic or Mild Symptoms of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT Kalbe Genexine Biologics (Industry)
Collaborators: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GXI7KGBio-001
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — efineptakin alfa

STUDY DESIGN:
Intervention Model Description: Double blinded phase 2 controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GX-I7 (Experimental): Patients randomised on experimental arm will receive GX-I7 drug
  Interventions: Drug: GX-I7
- GX-I7 vehicle (Placebo Comparator): Patients randomised on comparator arm will receive placebo
  Interventions: Drug: GX-I7

INTERVENTIONS:
Drug: GX-I7 — Recombinant human interleukin-7 hybrid Fc
  Other Names: Efineptakin alfa NT-I7; rhIL-7-hyFc; NT-I7; TJ107

SUMMARY:
This is a Phase 2 prospective, randomized, placebo-controlled, double-blinded, parallel group, single administration, multi-center study to assess the safety and efficacy of efineptakin alfa single treatment compared to placebo in elderly participants (adults ≥50years) with asymptomatic or mild COVID-19

DETAILED DESCRIPTION:
The study consists of 2 parts:

Part I - to identify the Recommended Phase 2 Dose (RP2D) compared to placebo in elderly participants (adults ≥50 years) with asymptomatic or mild COVID-19. These patients will be treated with 120 and 240 µg/kg efineptakin alfa, given on Day 1 (Baseline), respectively. The study will evaluate the safety, tolerability, and pharmacodynamics variable (ALC) of efineptakin alfa against COVID-19.

Part II - to assess the safety and efficacy of efineptakin alfa single treatment compared to placebo in elderly participants with asymptomatic or mild COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 50 years and above at the time of consent
2. Subjects who have been confirmed to be COVID-19 corresponding to asymptomatic case or mild cases of severity categorization classified by FDA through authorized molecular saliva-based test or polymerase chain reaction (PCR) test and who can be available to be administered within 7 days from the onset of any symptoms.
3. Patients who provide a voluntarily consent to participate in the study and sign the consent form in his/her own handwriting.
4. Female patients of childbearing potential (including female received a tubal ligation) should be prove negative pregnancy through pregnancy test before 24 hours of the IP administration, and must be willing to maintain abstinence (restraint sexual relationships) or use an adequate method of contraception at least 90 days after the IP administration.
5. Male patients must be willing to maintain abstinence (restraint sexual relationships) or use of adequate contraception method, and not to donate sperm. Men with childbearing or pregnant female spouses should maintain abstinence or use condoms at least 90 days after the IP administration to avoid exposure to embryos
6. Patients who agree for the hospitalisation (however, the hospitalisation will be performed only if needed)

Exclusion Criteria:

1. Patients who are unable to follow clinical and follow-up procedures
2. Patients with symptoms of moderate or higher in the severity classification presented by FDA have evidence of lower respiratory tract infection in their imaging findings or need supplemental oxygen therapy or mechanical respiration (ie, non-invasive ventilation, invasive mechanical ventilation, extracorporeal membrane oxygenation, etc)
3. Patients who have clinically significant cardiovascular diseases such as myocardial infarction, unstable arrhythmia and/or unstable angina within 3 months
4. Patients who have uncontrolled type II diabetes mellitus (despite the proper use of the drug, if fasting blood sugar level is not controlled to be more than 200 mg/dL)
5. If the principal investigator determines that patients are ineligible or difficult to follow the protocol due to evidence of severe or unregulated systemic diseases, uncontrolled hypertension (despite the proper use of the drug, if the blood pressure is not controlled to be lower than 150/90 mmHg), and active bleeding tendency
6. Patients who are known to be HIV positive
7. Patients who are known to be B-type, or C-type hepatitis-positive carrier
8. Patients who are pregnant or breastfeeding
9. Patients suspected of or identified with a malignant tumor or have a history of tumors within the past 5 years
10. Patients with the infectious diseases such as bacteremia or severe pneumonia requiring active treatment within four weeks prior to the IP administration
11. Patients with immunodeficiency or autoimmune diseases that can be exacerbated through immunotherapy at present
12. Patients who have previously received an allogeneic marrow transplantation or solid organ transplantation
13. Patients who are currently taking other drugs such as immunosuppressants that may affect the results of the study
14. Patients who have severe allergy for humanized antibodies or fusion proteins, anaphylaxis, or other hypersensitivity
15. Patients who have received other IP administration while participating in another clinical trial within 30 days prior to the IP administration for this study (However, biological preparation shall be applied to 60 days and even longer period can be applied considering the half-life) -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Dose finding | 9 weeks
  MTD and RP2D based on safety profiles
Absolute lymphocyte count (ALC) | 9 weeks
  The change of absolute lymphocyte count from baseline

SECONDARY OUTCOMES:
Treatment related Adverse Events | 10 weeks
  The proportion of participants with treatment emergent adverse events
Status of COVID-19 infection | 9 weeks
  Decrease of viral shedding identified with nasopharyngeal swab specimen by RT-PCR test
To evaluate the efficacy of GX-I7 in patients with COVID-19 | 9 weeks
  The proportion of participants who have progressed to moderate or severe or critical illness
Improvement in clinical parameters | 9 weeks
  Time to clinical improvement: clinical improvement is defined as a ≥ 2-point improvement in clinical status (8-point ordinal scale) from Day 1 (baseline)
Assess in improvement in clinical parameters | 9 weeks
  Time to ≥ 1-point improvement (days) from Day 1 (baseline) in terms of clinical status

OTHER OUTCOMES:
Immune repertoire in the study population | 9 weeks
  Changes of the rate of different immune cell types (i.e, effector/ memory T cell) and regulatory T cell (i.e, Tregs) in the blood after a single efineptakin alfa treatment, if possible

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Mitra Keluarga Kelapa Gading, Jakarta Pusat
  - Mitra Keluarga Kemayoran, Jakarta Pusat

IPD SHARING:
Plan to Share IPD: No